CLINICAL TRIAL: NCT04206787
Title: Real-world Study on Afatinib as First-line Treatment in Patients With Epidermal Growth Factor Receptor (EGFR) Mutation-positive Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: The Study Observes Afatinib as First-line Treatment in Patients With Epidermal Growth Factor Receptor (EGFR) Mutation-positive Advanced Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200-0318
Record Dates: First submitted 2019-12-11; First posted 2019-12-20 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Non-squamous, Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Afatinib-treated patients: Chinese patients with epidermal growth factor receptor (EGFR) mutation-positive advanced non-small cell lung cancer who initiated afatinib as first-line treatment. Patients received either 30 milligrams (mg) or 40 mg tablet of afatinib once daily as indicated in the approved label for the drug or any other subsequent therapy.
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — drug
  Other Names: Giotrif®

SUMMARY:
This study aims to observe the sequential strategy with afatinib as first-line treatment and to find the optimal treatment strategy for long-term chemotherapy-free regimens in Chinese patients with EGFR-mutated advanced NSCLC. Furthermore, this study can also assess the effectiveness and safety of afatinib as first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with locally advanced or metastatic NSCLC with EGFR sensitive mutation positive
* Patients who will initiate afatinib as first-line treatment for EGFR mutation-positive NSCLC
* Male and female patients with age ≥18 years
* Written informed consent per local regulatory requirement

Exclusion Criteria:

* Patients who have received previous systemic therapy (previous adjuvant or neoadjuvant therapies are permitted)
* Patients with symptomatic brain metastases (patients with brain metastases, who were previously treated, are eligible provided they have asymptomatic brain metastasis for at least 4 weeks on stable doses of medication) at the start of afatinib treatment
* Patients with concurrent participation in an interventional oncology clinical trial during the first-line treatment phase or within the last 30 days prior to the first-line treatment phase. If patients join another interventional study during the period of second-line treatment or later-line treatment, this patient should not be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be enrolled in this study and will receive afatinib (first-line) and subsequent treatment (second-line) of either 3rd generation EGFR TKI or other treatments
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Peking Union Medical College Hospital, Beijing
  - West China Hospital, Chengdu
  - The First Afiliated Hospital, Sun Yet-sen University, Guangzhou
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Hainan Cancer Hospital, Haikou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - China Shenyang Chest Hospital, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - The First Affiliated Hospital of Zhengzhou Unviersity, Zhengzhou
  - Zhongshan People's Hospital, Zhongshan

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-interventional, prospective, multicentre study based on real-world data of Chinese EGFR-mutated non-small cell-lung cancer (NSCLC) patients treated with afatinib as first-line treatment and receive subsequent therapy.
Pre-assignment Details: Only subjects that met all inclusion and none of the exclusion criteria were included. Patients were followed until death, lost to follow-up, withdraw from the study, or end of the study for other reasons, whichever came first and no later than 22-Dec-2023.
Period: Overall Study
Arm/Group | Afatinib-treated Patients
Started | 72
Treated | 72
Completed | 26
Not Completed | 46
Not completed — Other than listed | 2
Not completed — Investigator decision | 1
Not completed — Death | 25
Not completed — Lost to Follow-up | 9
Not completed — Withdrawal of consent | 9

BASELINE CHARACTERISTICS:
Population: Treated set: all patients who were dispensed medication and were documented to have taken at least one dose of first-line treatment afatinib.
Arm/Group | Afatinib-treated Patients
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 71
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Time on Treatment of Afatinib as First-line Therapy in Advanced Non-small Cell Lung Cancer Patients With Epidermal Growth Factor Receptor (EGFR) Mutation
Description: Time on Treatment (TOT) is defined as the median time a patient is under first-line afatinib treatment before being treated with third generation EGFR tyrosine kinase inhibitors (TKI) or other subsequent treatment, starting from the first dose of afatinib treatment until the last first-line dose or death by any cause, whichever comes first. Patients that were lost to follow up, withdrew before the end of study or received first-line afatinib at the end of the study were censored at the time of last known contact of first line afatinib.
  The median TOT was calculated using the Kaplan Mayer method and the 90% confidence interval was calculated using the Brookmeyer-Crowley method.
Time Frame: From first afatinib administration until last first-line afatinib administration, censoring date or death. Up to approximately 40 months.
Population: as for baseline characteristics
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Afatinib-treated Patients
Number analyzed (Participants) | 72
Months | 14.4 [11.27 to 18.07]

2. Secondary Outcome: Overall Survival (OS) From the Start of Afatinib Until the End of Study, Date of Death, Patient Withdrawal or Loss to Follow-up
Description: Overall survival (OS) is defined as the time from the start of afatinib until death for any reason. Subjects who have not died at the time of the statistical analysis were censored at the time they had the last known afatinib contact.
  The median survival time was calculated using the Kaplan Mayer method and the 90% confidence interval was calculated using the Brookmeyer-Crowley method. The median OS was not estimable due to the limited number of death events.
Time Frame: From first afatinib administration until death, or censoring date. Up to approximately 41 months.
Population: as for baseline characteristics
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Afatinib-treated Patients
Number analyzed (Participants) | 72
Months | NA [28.32 to NA] — Not estimable due to limited number of death events.

3. Secondary Outcome: Objective Response Rate (ORR) According to Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 by Investigator Review With Afatinib in First-line Treatment
Description: The objective response rate (ORR) is defined as the percentage of subjects treated with first-line afatinib with best overall response of complete response (CR), defined by the disappearance of all target lesions, and partial response (PR), defined by a decrease of at least 30% in the sum of the diameter of target lesions taking the baseline sum diameters as reference. The tumor response was evaluated by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
  The Clopper-Pearson method was used to provide an estimation of the ORR with 95% confidence interval.
Time Frame: From first afatinib administration until earliest RECIST progression (progressive disease (PD) or death) or the last evaluable assessment in the absence of RECIST progression (PD or death). Up to approximately 40 months.
Population: Treated set: all patients who were dispensed medication and were documented to have taken at least one dose of first-line treatment afatinib. Patients without tumor assessment data were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib-treated Patients
Number analyzed (Participants) | 67
Percentage of participants | 62.7 [50.01 to 74.20]

4. Secondary Outcome: Number of Patients With Any Adverse Event (AE)
Description: Number of patients treated with first-line afatinib with any adverse event.
Time Frame: From signing the informed consent form until 30 days after last dose of afatinib. Up to approximately 43 months.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib-treated Patients
Number analyzed (Participants) | 72
Participants | 68

5. Secondary Outcome: Number of Patients With Treatment-emergent Serious Adverse Events (SAE)
Description: Number of patients treated with first-line afatinib with treatment emergent serious adverse events (SAEs). SAEs are untoward medical occurrences that result in death, are life threatening, require inpatient hospitalisation, require prolongation of existing hospitalisation, result in persistent or significant disability/incapacity, result in a congenital anomaly/birth defect, or are deemed serious for any other medically important reason.
Time Frame: From first afatinib administration to 30 days after last dose of afatinib. Up to approximately 41 months.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib-treated Patients
Number analyzed (Participants) | 72
Participants | 10

6. Secondary Outcome: Number of Patients With Any Afatinib-related Adverse Events (AE)
Description: Number of patients treated with first-line afatinib with any adverse event associated with the use of afatinib.
Time Frame: From first afatinib administration to 30 days after last dose of afatinib. Up to approximately 41 months.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Afatinib-treated Patients
Number analyzed (Participants) | 72
Participants | 63

ADVERSE EVENTS:
Time Frame: All-cause mortality: From first afatinib administration until individual end of study. Up to approximately 43 months. Treatment-emergent adverse event reporting: From first afatinib administration until last afatinib administration plus 30 days residual effect period (REP). Up to approximately 41 months.
Description: Treated set: all patients who were dispensed medication and were documented to have taken at least one dose of first-line treatment afatinib.
Arm/Group | Afatinib-treated Patients
All-Cause Mortality (participants affected / at risk) | 25/72
Serious Adverse Events (participants affected / at risk) | 10/72
Other Adverse Events (participants affected / at risk) | 65/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib-treated Patients (N=72)
Nausea (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death (General disorders) | 1
COVID-19 (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib-treated Patients (N=72)
Anaemia (Blood and lymphatic system disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 53
Mouth ulceration (Gastrointestinal disorders) | 34
Pyrexia (General disorders) | 4
Hepatic function abnormal (Hepatobiliary disorders) | 6
Paronychia (Infections and infestations) | 23
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 7
Headache (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT04206787/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT04206787/SAP_001.pdf